CLINICAL TRIAL: NCT04490694
Title: TACE Combined With Lenvatinib for Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-151R
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Transarterial Chemoembolization; lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE Combined with Lenvatinib (Experimental)
  Interventions: Drug: Lenvatinib; Procedure: TACE

INTERVENTIONS:
Drug: Lenvatinib — Intervention Description：lenvatinib will be administered daily (for patients <60kg, lenvatinib 8mg bid po for patients ≥60kg, lenvatinib 12mg bid po) until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Other Names: Lenvatinib treatment
Procedure: TACE — Patients will be treated with TACE 2-4 weeks after randomization: the blood supply of the tumor will be evaluated by transradial / femoral artery approach, microcatheter will be inserted into the tumor feeding artery, and lipiodol plus epirubicin emulsifier will be injected (40mg epirubicin will be added to each 10ml lipiodol, the total amount should less than 20ml, epirubicin 40-60mg). Gelatin sponge particles / microspheres are used to strengthen embolization. Blood biochemical examination will be performed within 1 week before TACE, 3 days after operation and 1 month after operation.
  Other Names: Transcatheter arterial chemoembolization

SUMMARY:
It is an exploratory clinical study aimed to evaluate the efficacy and safety of TACE combined with Lenvatinib in the treatment of patients with BCLC stage B and C HCC.Treatment will continue until the death or intolerable toxicity or patients withdrawal of consent,and the target sample size is 54 individuals.

DETAILED DESCRIPTION:
This is a prospective, single-center and single-arm exploratory clinical study designed to evaluate the efficacy and safety of TACE combined with Lenvatinib in the treatment of patients with BCLC stage B and C hepatocellular carcinoma.Treatment will continue until the death or intolerable toxicity or patients withdrawal of consent,and the target sample size is 54 individuals.

ELIGIBILITY:
Inclusion Criteria:

- 1. Histopathologically or clinically confirmed unresectable hepatocellular carcinoma.

2. Age ≥ 18 years at time of study entry. 3. Child-Pugh scores <7. 4. Performance status (PS) ≤ 2 (ECOG scale). 5. BCLC stage B, some patients in stage C (Vp2-3). 6. The patient and/or his family agreed to join the clinical trial and sign the informed consent form.

Exclusion Criteria:

* 1. Have received TACE or other local treatment for liver cancer (except bridged liver transplantation).

  2. Main portal vein tumor thrombus or complicated with extrahepatic metastasis. 3. Tumor burden≥70% , diffuse liver cancer or tumor is not suitable for mRECIST standard evaluation.

  4. Have received systemic chemotherapy, sorafinib or other targeted therapy or immunotherapy.

  5. Estimated life expectancy of <3 months. 6. There is a significant decrease in white blood cells and platelets in peripheral blood, severe coagulation dysfunction and can not be corrected：the neutrophil<1.5×109/L, PLT<50×109/L. The INR>2.3.

  7. Renal dysfunction：serum creatinine (SCR) >176.8 μmol/L（2 mg/dL）or creatinine clearance rate (Ccr) <30 mL/min.

  8. Serious heart, lung, brain or other important organ diseases. 9. Pregnant or lactating women. 10. cannot cooperate with TACE operation and sign informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to progression（TTP） | 2 years
  The time from the beginning of randomization to the tumor progression of the patient
Objective remission rate（ORR） | 2 years
  ORR according to modified RECIST for Hepatocellular Carcinoma

SECONDARY OUTCOMES:
Adverse Events | 2 years
  Adverse event (AE)、Treatment emergent adverse event(TEAE)、Serious adverse event (SAE)
Overall survival | 5 years
  the survival time after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zhiping Yan, M.D., Principal Investigator — Fudan University
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University., Shanghai, Shanghai Municipality, China